CLINICAL TRIAL: NCT02375568
Title: Large-scale ex Vivo Expansion and Characterization of Synovial Membrane Mesenchymal Stem Cells (SM-MSC) and Infrapatellar Fat Pad Mesenchymal Stem Cells (IF-MSC) for Clinical Application
Brief Title: Large-scale Expansion and Characterization of Mesenchymal Stem Cells for Clinical Application
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chin-Hung Chang (Other)
Collaborators: EMO Biomedicine Corporation (Industry)
Responsible Party: Sponsor-Investigator, Chin-Hung Chang, MD. PhD., Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Other Study IDs: 201405EMO
Record Dates: First submitted 2015-02-10; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Knee Injuries
Keywords: mesenchymal stem cells
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 103024-F: For patients who have an operation of total knee replacement, two removed tissues (synovial membrane and infrapatellar fat pad) will be collected for mesenchymal stem cell isolation.
  Interventions: Other: 103024-F

INTERVENTIONS:
Other: 103024-F — mesenchymal stem cell isolation

SUMMARY:
According to many recent research, mesenchymal stem cells (MSC) isolated from synovial membrane and infrapatellar fat pad have higher ex vivo proliferation capacity, multipotency and ability to undergo chondrogenesis.

Based on this concept, the investigators plan to get two removed tissues (synovial membrane and infrapatellar fat pad) from patients who have an operation of total knee replacement. The investigators are going to isolate and expand MSC from these two tissues respectively, and then compare the chondrogenesis ability for clinical application. In the other hand, the investigators plan to build techniques and procedures which comply with "Good Tissue Practices (GTP)"

ELIGIBILITY:
Inclusion Criteria:

Patient who have an total knee replacement surgery

Exclusion Criteria:

Patient who don't sign the agreement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who have an total knee replacement surgery
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Cell viability ratio of synovial membrane MSC and infrapatellar fat pad MSC from the first to the tenth cell passage | 6 months
Doubling time of synovial membrane MSC and infrapatellar fat pad MSC from the first to the tenth cell passage | 6 months
Percentage expression of cluster differentiation 90,105, 34, 45 surface markers of synovial membrane MSC and infrapatellar fat pad MSC from the first to the tenth cell passage | 6 months

SECONDARY OUTCOMES:
Alcian blue staining of synovial membrane MSC and infrapatellar fat pad MSC | 6 months
Tyep II collagen and aggrecan gene expression of synovial membrane MSC and infrapatellar fat pad MSC | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Pan-Ciao, Taipei, Taiwan